CLINICAL TRIAL: NCT06768710
Title: PECARN Versus NICE Guidelines for Pediatric Head Trauma in Emergency Department in Assuit and Sohag University Hospitals
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Noha Badran Abdelmawgoud, resident doctor at Emergency medicine, Sohag University, Sohag University
Other Study IDs: PECARN vs NICE head trauma
Record Dates: First submitted 2024-12-22; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Head Trauma
Keywords: NICE Guidelines; PECARN Guidelines
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- head trauma patients: patients less than 16 years old with head trauma indicated for CT brain according to current clinical practice

SUMMARY:
the safety and validity of the PECARN with 100% sensitivity in both age groups in identifying patients with ciTBI and theoretically in reducing performed CT scans by 29%. Therefore, in patients classified in the low-risk category, it is a duty not to expose the child to ionizing radiation.

the NICE criteria can minimize the number of CT scans conducted while maintaining a fair sensitivity for identifying patients with TBI and those requiring neurosurgical intervention the sensitivity of the intracranial damage NICE criteria was 93% for early presenters.

This study is conducted to detect which guidelines can be followed to detect all intracranial lesions with minimizing the number of unnecessary CT scans.

the aim of the study is to evaluate safety and efficacy (sensitivity and specificity) of PECARN and NICE guidelines for detection of traumatic brain injury as compared to current clinical practice in emergency setting and Detection of intracranial findings on CT brain and detection of lesions that need neurosurgical intervention.

Significance of the study:

DETAILED DESCRIPTION:
Head trauma in children is one of the most common causes for emergency department (ED) visits. Most head trauma incidents in children visiting the ED are minor; however, identifying those patients who have clinically important traumatic brain injury (ciTBI) is challenging.

A cranial computed tomography (CT) scan is the standard diagnostic test and is widely used all over the world. Although cranial CT scans are useful for definitive diagnosis, potential cancer risks exist associated with ionizing radiation, particularly in children, who are more radiosensitive than adults.

Head trauma prediction rules have been derived for supporting phyiscians to improve accuracy in decision-making and to minimize the use of potentially harmful CT scans. The Pediatric Emergency Care Applied Research Network (PECARN) developed two age-based head trauma prediction rules to identify children with very low risk of ciTBI who do not require cranial CT scans .

The PECARN rule was statistically derived to identify children at very low risk of ciTBI for whom a CT scan could safely be avoided based on the absence of predictor variables. In the presence of predictor variables, the algorithm stratifies the management of children into an intermediate-risk or high-risk group based on the risk of ciTBI. Children at high risk are recommended to have a CT scan as the risk of ciTBI outweighs the risks associated with radiation exposure.

NICE guideline: This guideline covers assessment and early management of head injury in infants, children, young people and adults. It aims to ensure that people have the right care for the severity of their head injury, including direct referral to specialist care if needed. This guideline has updated some of the terminology used in relation to safeguarding people under 16. according to algorithm 2 page8.

ELIGIBILITY:
Inclusion Criteria:

* All patients less than 16 years old with head trauma indicated for CT brain according to current clinical practice.

Exclusion Criteria:

-Patients unstable to had a CT scan.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients less than 16 years old with head trauma indicated for CT brain according to current clinical practice
Sampling Method: Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
the accuracy of PECARN guidelines | 30 day
  evaluate the accuracy of PECARN guidelines for detection of traumatic brain injury
the accuracy of NICE guidelines | 30 day
  evaluate the accuracy of NICE guidelines for detection of traumatic brain injury

IPD SHARING:
Plan to Share IPD: Undecided